CLINICAL TRIAL: NCT07288463
Title: Hearing Loss and Genetic Risks for Dementia
Brief Title: Hearing Loss and Genetic Risks for Alzheimer's Disease and Related Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Janet Choi, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APP-25-05793
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss, Adult-Onset; Dementia
MeSH Terms: conditions — Hearing Loss; Dementia | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate Intervention (Experimental): Immediate Intervention: 4-month of OTC hearing aid use
  Interventions: Device: Over-The-Counter (OTC) hearing aid
- Waitlist control (Active Comparator): Waitlist control: Basic patient education on hearing loss without OTC hearing aid for 2 months, followed by 4 months of OTC hearing aid use
  Interventions: Device: Over-The-Counter (OTC) hearing aid

INTERVENTIONS:
Device: Over-The-Counter (OTC) hearing aid — Over-The-Counter (OTC) hearing aid

SUMMARY:
Hearing loss is a prevalent and modifiable risk factor for cognitive decline and dementia in older adults, yet access to hearing care remains limited. Over-the-counter (OTC) hearing aids represent a promising and scalable strategy to expand access, particularly for individuals at elevated risk for dementia who may benefit most from earlier intervention. This pilot study aims to evaluate the feasibility and acceptability of OTC hearing aid use among older adults at increased risk for dementia. Participants aged ≥50 years will undergo standardized hearing screening to identify bilateral, mild-to-moderate hearing loss. Eligible participants will be randomized to one of two sequences: (1) immediate intervention: 4-mo using OTC hearing aids or (2) waitlist control: 2-mo without devices followed by an additional 4-mo using OTC hearing aids. Feasibility outcomes include study enrollment and retention, protocol adherence, and average daily device use determined by data-logging. Acceptability outcomes will be assessed using the International Outcome Inventory for Hearing Aids (IOI-HA), device satisfaction ratings, and participant intention to continue hearing-aid use. Hearing outcomes include validated questionnaires on hearing and listenign efforts. Findings will inform the design of larger trials aimed at improving access to hearing care and promoting cognitive health in high-risk older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 50 years
* APOE ε4 carriers
* Bilateral mild to moderate sensorineural hearing loss
* No current use of hearing aids or cochlear implants
* No diagnosis of dementia and able to provide informed consent
* Able to complete questionnaires and follow instructions in English
* Willing and able to comply with study procedures, follow-up visits, and hearing-aid use

Exclusion Criteria:

* Clinical diagnosis of dementia
* Severe or profound hearing loss
* Self-reported congenital hearing loss
* Absence of an ear canal due to medical conditions or prior surgical procedures
* unwillingness to wear OTC hearing aids regularly (>=4 hours/day)
* medical contraindication to use hearing aids (e.g., actively draining ear)
* Known retrocochlear pathology
* Severe uncorrected visual impairment or significant manual dexterity limitations that prevent handling the device

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility- Proportion of enrolled participants who complete all study periods | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility- Proportion of enrolled participants who complete all study periods
Feasibility - Enrollment rate (% eligible who consent) | Baseline
  Feasibility - Enrollment rate (% eligible who consent)
Feasibility - Study visit completion rate (% of planned visits completed) | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Study visit completion rate (% of planned visits completed)
Feasibility - Frequency of device troubleshooting encounters | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Frequency of device troubleshooting encounters
Feasibility - Percentage achieving >= 4hours/day of objective wear time | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Percentage achieving >= 4hours/day of objective wear time
Feasibility - Hearing aid use adherence (mean daily wear time from data-logging) | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Hearing aid use adherence (mean daily wear time from data-logging)
Feasibility - Protocol adherence rate (% completing scheduled assessments) | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Protocol adherence rate (% completing scheduled assessments)
Feasibility - Retention rate (% completing follow-up visits) | Baseline, 2-months, 4-months, and 6-months follow up
  Feasibility - Retention rate (% completing follow-up visits)
Acceptability - International Outcome Inventory for Hearing Aids | Baseline, 2-months, 4-months, and 6-months follow up
  International Outcome Inventory for Hearing Aids
Acceptability - Intention to continue use after study completion | Baseline, 2-months, 4-months, and 6-months follow up
  Acceptability - Intention to continue use after study completion

SECONDARY OUTCOMES:
Hearing Handicap Inventory - Screening Version | Baseline, at the end of period 1 (4-week from baseline), at the end of period 2 (8-week from baseline)
  Hearing Handicap Inventory - Screening Version
Vanderbilt fatigue scale | Baseline, 2-months, 4-months, and 6-months follow up
  Listeing-related fatigue: Vanderbilt fatigue scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, individual participant data (IPD) will not be shared. Because this is a small feasibility pilot study involving a high-risk population, and the primary study outcomes are feasibility and acceptability metrics rather than clinical endpoints, we do not anticipate that sharing individual-level data would provide meaningful scientific value.